CLINICAL TRIAL: NCT05492721
Title: Comparing Tissue Adhesives in Port Site Closure: A Randomized Controlled Trial
Brief Title: Comparing Tissue Adhesives in Port Site Closure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Julie Holihan, Assistant Professor of Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-22-0143
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dermatitis, Contact
Keywords: GLUE; SURGICAL GLUE; DERMABOND; DERMATITIS
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis

STUDY DESIGN:
Intervention Model Description: Each subject will have both glue types and serve as their own control
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor does not know which glue was used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dermabond (Active Comparator): Dermabond over incisions
  Interventions: Device: 2-Octylcyanoacrylate
- Swiftset (Active Comparator): Swiftset over incisions
  Interventions: Device: N-butyl-2-cyanoacrylate

INTERVENTIONS:
Device: 2-Octylcyanoacrylate — Incisions on left will have one glue and on right will have the other glue
  Other Names: Dermabond
  Arms: Dermabond
Device: N-butyl-2-cyanoacrylate — Incisions on left will have one glue and on right will have the other glue
  Other Names: Swiftset
  Arms: Swiftset

SUMMARY:
This is a multi-center randomized controlled trial to evaluate two different methods of reinforcing surgical port site closure: 2-Octylcyanoacrylate and n-butyl-2-cyanoacrylate.

DETAILED DESCRIPTION:
Study Design

This is a multi-center randomized controlled trial to evaluate two different methods of reinforcing surgical port site closure: 2-Octylcyanoacrylate and n-butyl-2-cyanoacrylate.

Methods

Inclusion Criteria All adult patients undergoing an elective laparoscopic or robotic abdominal surgery with the Minimally Invasive Surgeons of Texas (MIST) either at Texas Medical Center or Sugar Land will be eligible.

Exclusion criteria

1. Patients unlikely to follow-up (live out of state, unable to be reached by phone or email)
2. Patients with a known allergy to 2-Octylcyanoacrylate or N-butyl-2-cyanoacrylate.

Treatment Groups Eligible patients will be approached by research staff either in clinic or in pre-operative holding for trial enrollment. Each patient will serve as their own control. Enrolled patients will have both surgical glue types used, one on each half of their abdomen. The side for each glue will be randomly assigned by the day of the month. On odd days, 2-Octylcyanoacrylate will go on the patient's left abdomen. On even days, 2-Octylcyanoacrylate will go on the patient's right abdomen. If there is an odd number of incisions, the extra incision will be included on the patient's left.

All incisions will be closed with Monocryl. Closed incisions will be covered with skin glue.

Outcome The primary outcome of this trial will be the proportion of patients with contact dermatitis within 6 weeks post-operative. A trained surgical clinician blinded to the treatment arms will collect outcomes at all follow up clinic visits in the first 6 weeks post-operative. Any skin reaction will be documented with photographs.

Secondary outcome will include the diameter of erythema around any skin reaction, or any wound dehiscence or surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* undergoing an elective laparoscopic or robotic abdominal surgery

Exclusion Criteria:

* Patients unlikely to follow-up (live out of state, unable to be reached by phone or email)
* Patients with a known allergy to 2-Octylcyanoacrylate or N-butyl-2-cyanoacrylate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
proportion of patients who develop contact dermatitis | 6 weeks
  erythema or rash around incisions

SECONDARY OUTCOMES:
mean diameter of erythema | 6 weeks
  mean diameter of erythema around incisions for those with contact dermatitis
proportion of patients with wound dehiscence | 6 weeks
  opening of incisions
proportion of patients with surgical site infection | 6 weeks
  CDC definition of surgical site infection

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No